CLINICAL TRIAL: NCT03110809
Title: The Effects of Capsinoids on Brown Adipose Tissue Recruitment and Activation in Obesity
Brief Title: The Effects of Capsinoids on Brown Adipose Tissue Activation in Obesity
Acronym: BATCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lisa Neff, Medical Doctor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SP0037287
Record Dates: First submitted 2017-03-20; First posted 2017-04-12 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Weight Loss
Keywords: obesity; brown; fat; weight; loss
MeSH Terms: conditions — Weight Loss; Obesity; Platelet Glycoprotein IV Deficiency; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAT Positive Placebo (Placebo Comparator): Participants will be confirmed positive for BAT activity, but on Placebo
  Interventions: Dietary Supplement: Placebo
- BAT Negative Placebo (Placebo Comparator): Participants will be confirmed negative for BAT activity, but on Placebo
  Interventions: Dietary Supplement: Placebo
- BAT Positive Capsinoid (Experimental): Participants will be confirmed positive for BAT activity, but taking Capsinoids. Capsinoids are a derivative of sweet peppers that may activate and recruit BAT.
  Interventions: Dietary Supplement: Capsinoid
- BAT Negative Capsinoid (Experimental): Participants will be confirmed negative for BAT activity, but taking Capsinoids. Capsinoids are a derivative of sweet peppers that may activate and recruit BAT.
  Interventions: Dietary Supplement: Capsinoid

INTERVENTIONS:
Dietary Supplement: Capsinoid — Capsinoids are nunpungent analogs of capsaicin that activate BAT by stimulating sensory neurons in the gastrointestinal tract. Chronic ingestion of capsinoids may stimulate the development or recruitment of new BAT from precursor stem cells within white adipose tissue depots.
  Arms: BAT Negative Capsinoid; BAT Positive Capsinoid
Dietary Supplement: Placebo — Placebo for capsinoid. Capsule contains no active ingredients.
  Arms: BAT Negative Placebo; BAT Positive Placebo

SUMMARY:
This research study is being done to determine whether taking a dietary supplement called capsinoids, derived from sweet peppers, can activate brown fat that is already present or even generate new brown fat in individuals with excess weight. Previous studies have suggested that chronic consumption of capsinoids may be able to generate new brown fat in thin individuals. Capsinoids may also have a small positive effect on metabolism (increased calorie-burning) and fat loss. The knowledge gained in this study may eventually lead to more treatment options for people with excess weight.

DETAILED DESCRIPTION:
Obesity has become an epidemic in the United States, affecting more than one-third of American adults and increasing the incidence of diabetes and other comorbidities. Weight loss elicits adaptive metabolic and hormonal changes, similar to those seen in starvation, which make maintenance of a reduced body weight more challenging. These changes include a decrease in energy expenditure that is larger than what would be expected on the basis of changes in body composition alone. In rodents, it has long been established that brown adipose tissue (BAT) is the primary site of adaptive thermogenesis or the modulation of energy expenditure and heat generation during cold exposure and overfeeding. Emerging data suggest that activated BAT may influence body weight, core body temperature, energy expenditure and blood sugar and fat metabolism in humans. Capsinoids are nunpungent analogs of capsaicin that activate BAT by stimulating sensory neurons in the gastrointestinal tract. Chronic ingestion of capsinoids may stimulate the development or recruitment of new BAT from precursor stem cells within white adipose tissue depots. The primary goal of the proposed study is to determine whether chronic ingestion of capsinoids can recruit BAT in obese individuals who lack it or merely activates BAT in those who already have it. Additional goals are to 1) ascertain whether common genetic variants influence the response to capsinoids, 2) determine the metabolic effects of chronic capsinoid ingestion and BAT activation in obesity without weight loss and 3) establish whether chronic capsinoid ingestion and BAT activation improve weight loss with a low calorie diet. 42 obese male volunteers, ages 18-50, will be recruited for a randomized, double-blind, placebo-controlled trial of capsinoid supplementation. The study will consist of two phases: the first in which subjects maintain their usual diet and activity level for 8 weeks, and the second in which subjects consume a low-calorie diet for 12 weeks. Subjects will be studied before and after each phase, including measurement of BAT, core body temperature, energy expenditure at rest, after cold exposure, and after a test meal, body composition, and blood sugar and insulin levels after a test meal. BAT will be characterized using Positron Emission Tomography/Magnetic Resonance (PET/MR) and Magnetic Resonance Imaging (MRI) techniques. If preliminary data are confirmed, BAT recruitment and activation through chronic capsinoid supplementation may emerge as a safe method to combat the adaptive changes in energy expenditure that are seen with weight loss in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* 18-50 years old.
* Non-smoking.
* Overweight/Obese (BMI 27-45).
* Generally healthy.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
MRI BAT activity maps | 22 weeks
  Develop multi-parametric MRI BAT activity maps by comparing MRI measurements at thermo-neutral, non-shivering thermogenesis and warm-up conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Neff, MD., MS., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No